CLINICAL TRIAL: NCT00085709
Title: A Phase III Study of the Addition of Gemtuzumab Ozogamicin (Mylotarg®) During Induction Therapy Versus Standard Induction With Daunomycin and Cytosine Arabinoside Followed by Consolidation and Subsequent Randomization to Post-Consolidation Therapy With Gemtuzumab Ozogamicin (Mylotarg®) or No Additional Therapy For Patients Under Age 61 With Previously Untreated De Novo Acute Myeloid Leukemia (AML)
Brief Title: S0106 Cytarabine and Daunorubicin w/ or w/o Gemtuzumab Followed By HD Cytarabine and Either Gemtuzumab or Nothing in de Novo AML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S0106; U10CA032102 (NIH); S0106 (Other: SWOG)
Record Dates: First submitted 2004-06-14; First posted 2004-06-16 (Estimated); Results first posted 2012-08-27 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute eosinophilic leukemia; adult acute basophilic leukemia; adult acute monocytic leukemia (M5b); adult acute erythroid leukemia (M6); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Eosinophilic, Acute; Leukemia, Basophilic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities | interventions — Gemtuzumab; Observation; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Post-consolidation GO (Experimental): Patients receive gemtuzumab ozogamicin IV over 2 hours on day 1. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemtuzumab ozogamicin
- Post-consolidation observation (Other): Patients receive no additional therapy. Patients are observed at days 30 and 60 after randomization.
  Interventions: Other: observation
- Induction 7+3 (Active Comparator): Standard induction regimen of 7 days of Ara-C (cytosine arabinoside) and 3 days of daunomycin
  Interventions: Drug: Cytosine arabinoside; Drug: Daunomycin
- Induction 7+3+GO (Active Comparator): Gemtuzumab (GO) added to the standard induction regimen of 7 days of Ara-C and 3 days of daunomycin
  Interventions: Drug: Cytosine arabinoside; Drug: Daunomycin

INTERVENTIONS:
Drug: gemtuzumab ozogamicin — Given IV, induction Arm1 6mg/m2 D4; post-consolidation 5mg/m2 3 doses >/= 28 days apart
  Other Names: mylotarg
  Arms: Post-consolidation GO
Other: observation — No treatment given
  Arms: Post-consolidation observation
Drug: Cytosine arabinoside — IV; induction Arms1/2 and reinduction 100 mg/m2/d days 1-7; consolidation 3gm/m2 q3hrs D1, 3, 5
  Other Names: Ara-C
  Arms: Induction 7+3; Induction 7+3+GO
Drug: Daunomycin — IV; induction Arm1 45mg/m2 D1-3; Arm2 and reinduction 60 mg/m2 D1-3;
  Other Names: daunorubicin
  Arms: Induction 7+3; Induction 7+3+GO

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cytarabine and daunorubicin, work in different ways to stop cancer cells from dividing so they stop growing and die. Monoclonal antibodies, such as gemtuzumab ozogamicin, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining chemotherapy with gemtuzumab ozogamicin may kill more cancer cells. It is not yet known whether induction therapy using cytarabine and daunorubicin is more effective with or without gemtuzumab ozogamicin or whether postconsolidation therapy using gemtuzumab ozogamicin is more effective than no additional therapy in treating de novo (first occurrence) acute myeloid leukemia.

PURPOSE: This randomized phase III trial is comparing two different regimens of chemotherapy and monoclonal antibody therapy to see how well they work in treating patients with previously untreated de novo acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare disease-free survival of patients with previously untreated de novo acute myeloid leukemia treated with induction therapy comprising cytarabine and daunorubicin with vs without gemtuzumab ozogamicin followed by consolidation therapy comprising high-dose cytarabine and post-consolidation therapy comprising gemtuzumab ozogamicin vs no additional therapy.
* Compare the complete remission rate in patients treated with these regimens.
* Compare the frequency and severity of the toxic effects of these regimens in these patients.

Other objectives (if funding allows):

* Determine the prognostic significance of CD33 expression on the response rate in patients receiving gemtuzumab ozogamicin.
* Determine the prognostic significance of FLT3 mutations in these patients before treatment with these regimens.
* Determine the prognostic significance of minimal residual disease in remission specimens from these patients treated with these regimens.
* Determine the prognostic significance of the flow cytometric detection of minimal residual disease in specimens collected from these patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified during induction therapy according to age (< 35 years vs ≥ 35 years) and during post-consolidation therapy according to preinduction cytogenetic risk group.

* Induction therapy: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive daunorubicin IV on days 1-3, cytarabine IV continuously on days 1-7, and gemtuzumab ozogamicin IV over 2 hours on day 4. Patients receive filgrastim (G-CSF) or sargramostim (GM-CSF) IV or subcutaneously once daily beginning on day 15 and continuing until blood counts recover.
  * Arm II: Patients receive daunorubicin, cytarabine, and G-CSF or GM-CSF as in arm I.

Patients in both arms undergo bone marrow aspiration and biopsy on day 14 (and on day 19, if applicable) and then proceed to reinduction therapy.

* Reinduction therapy: Patients receive daunorubicin IV on days 1-3 and cytarabine IV continuously on days 1-7. Patients also receive G-CSF or GM-CSF as in induction therapy.

Patients who achieve A1 bone marrow, B1 peripheral blood, and C1 extramedullary disease status proceed to consolidation therapy.

* Consolidation therapy: Patients receive high-dose cytarabine IV over 3 hours twice daily on days 1, 3, and 5. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients who maintain A1 bone marrow, B1 peripheral blood, and C1 extramedullary disease status after consolidation therapy proceed to post-consolidation therapy.

* Post-consolidation therapy: Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive gemtuzumab ozogamicin IV over 2 hours on day 1. Treatment repeats every 28 days for 3 courses in the absence of disease progression or unacceptable toxicity.
  * Arm II: Patients receive no additional therapy. Patients are observed at days 30 and 60 after randomization.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 684 patients (342 per treatment arm) will be accrued for this study within 4.5-5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically confirmed acute myeloid leukemia (AML) by bone marrow aspiration and biopsy* within the past 14 days

  * No M3 disease NOTE: *Patients with marked leukocytosis may be registered before the availability of biopsy results if the absolute blast count is ≥ 100,000 cells/µL
* No blastic transformation of chronic myelogenous leukemia
* No pre-existing hematologic disorder evolving to AML (e.g., myelodysplasia or secondary leukemia)

PATIENT CHARACTERISTICS:

Age

* 18 to 60

Performance status

* Zubrod 0-3

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* No known hepatitis B or C infection
* No known liver disease

Renal

* Not specified

Cardiovascular

* LVEF ≥ 50% by MUGA or echocardiogram
* No unstable cardiac arrhythmias
* No unstable angina

Other

* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior systemic chemotherapy

  * Prior hydroxyurea to control high cell counts allowed
* No more than 1 prior dose of intrathecal chemotherapy for acute leukemia
* Concurrent intrathecal chemotherapy allowed during induction therapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 637 (Actual)
Dates: Start 2004-07; Primary Completion 2010-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen H. Petersdorf, MD, Study Chair — Seattle Cancer Care Alliance
Locations (279):
- United States (255):
  - Providence Cancer Center, Anchorage, Alaska
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Sutter Solano Medical Center, Vallejo, California
  - Center for Cancer Care and Research at Watson Clinic, LLP, Lakeland, Florida
  - Phoebe Cancer Center at Phoebe Putney Memorial Hospital, Albany, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (16):
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Moncton Hospital, Moncton, New Brunswick
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Charles Lemoyne, Greenfield Park, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- Sweden (8):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital - Huddinge, Huddinge
  - University Hospital of Linkoping, Linköping
  - Lund University Hospital, Lund
  - Orebro University Hospital, Örebro
  - Karolinska University Hospital - Solna, Stockholm
  - Sundsvall Hospital, Sundsvalls
  - Uppsala University Hospital, Uppsala

REFERENCES:
- [Derived] Dillon LW, Higgins J, Nasif H, Othus M, Beppu L, Smith TH, Schmidt E, Valentine Iii CC, Salk JJ, Wood BL, Erba HP, Radich JP, Hourigan CS. Quantification of measurable residual disease using duplex sequencing in adults with acute myeloid leukemia. Haematologica. 2024 Feb 1;109(2):401-410. doi: 10.3324/haematol.2023.283520. PMID 37534515
- [Derived] Zarnegar-Lumley S, Alonzo TA, Gerbing RB, Othus M, Sun Z, Ries RE, Wang J, Leonti A, Kutny MA, Ostronoff F, Radich JP, Appelbaum FR, Pogosova-Agadjanyan EL, O'Dwyer K, Tallman MS, Litzow M, Atallah E, Cooper TM, Aplenc RA, Abdel-Wahab O, Gamis AS, Luger S, Erba H, Levine R, Kolb EA, Stirewalt DL, Meshinchi S, Tarlock K. Characteristics and prognostic impact of IDH mutations in AML: a COG, SWOG, and ECOG analysis. Blood Adv. 2023 Oct 10;7(19):5941-5953. doi: 10.1182/bloodadvances.2022008282. PMID 37267439
- [Derived] Medeiros BC, Othus M, Fang M, Appelbaum FR, Erba HP. Cytogenetic heterogeneity negatively impacts outcomes in patients with acute myeloid leukemia. Haematologica. 2015 Mar;100(3):331-5. doi: 10.3324/haematol.2014.117267. Epub 2014 Dec 19. PMID 25527568
- [Derived] Medeiros BC, Othus M, Estey EH, Fang M, Appelbaum FR. Unsuccessful diagnostic cytogenetic analysis is a poor prognostic feature in acute myeloid leukaemia. Br J Haematol. 2014 Jan;164(2):245-50. doi: 10.1111/bjh.12625. Epub 2013 Oct 28. PMID 24383844
- [Derived] Petersdorf SH, Kopecky KJ, Slovak M, Willman C, Nevill T, Brandwein J, Larson RA, Erba HP, Stiff PJ, Stuart RK, Walter RB, Tallman MS, Stenke L, Appelbaum FR. A phase 3 study of gemtuzumab ozogamicin during induction and postconsolidation therapy in younger patients with acute myeloid leukemia. Blood. 2013 Jun 13;121(24):4854-60. doi: 10.1182/blood-2013-01-466706. Epub 2013 Apr 16. PMID 23591789

RESULTS

PARTICIPANT FLOW:
Groups:
- Ara-C+Daunomycin+Mylotarg: Gemtuzumab (GO) added to the standard induction regimen of 7 days of Ara-C (cytosine arabinoside)and 3 days of daunomycin
- ARA-C+Daunomycin: Standard induction regimen of 7 days of Ara-C (cytosine arabinoside)and 3 days of daunomycin
Period: Overall Study
Arm/Group | Ara-C+Daunomycin+Mylotarg | ARA-C+Daunomycin
Started | 317 | 320
Eligible | 298 | 301
Eligible and Did Not Withdraw Consent | 296 | 300
Completed | 264 | 270
Not Completed | 53 | 50
Not completed — Adverse Event | 8 | 0
Not completed — Death | 8 | 2
Not completed — Refusal unrelated to adverse events | 1 | 2
Not completed — Progression | 3 | 4
Not completed — Not protocol specified | 12 | 22
Not completed — Not eligible | 19 | 19
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ara-C+Daunomycin+Mylotarg: Ara-C+Daunomycin+Mylotarg
- ARA-C+Daunomycin: ARA-C+Daunomycin
- Total: Total of all reporting groups
Arm/Group | Ara-C+Daunomycin+Mylotarg | ARA-C+Daunomycin | Total
Number analyzed (Participants) | 296 | 300 | 596
Age, Continuous [Median (Full Range); unit: years] | 47 [18 to 60] | 48 [18 to 60] | 47 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 148 | 283
  Male | 161 | 152 | 313

OUTCOME MEASURES:

1. Primary Outcome: 2-year Disease-free Survival (DFS)
Description: Measured from data of randomization to post-consolidation therapy until relapse from complete response or death from any cause, with observations censored at the date of last contact for patients last known to be alive without report of relapse.
Time Frame: After completing any treatment, every 6 months for 2 years, than annually for years 3-5
Population: Eligible patients who completed induction and consolidation therapy
Measure: Number (95% Confidence Interval); unit: Percentage of population
Groups:
- Post-consolidation GO: For patients who remain in CR without relapse, patients may receive up to 3 doses of G.O. 28 days apart.
- Post-consolidation Observation: Patients did not receive any post-consolidation therapy
Arm/Group | Post-consolidation GO | Post-consolidation Observation
Number analyzed (Participants) | 84 | 84
Percentage of population | 39 [27 to 51] | 50 [38 to 62]
Statistical Analysis 1: Comparison: Post-consolidation GO vs Post-consolidation Observation; Interim futility analysis of the alternative hypothesis for disease-free survival. The design specified a hazard ratio of (observation: GO) of 1.5; Test type: Superiority or Other; p < 0.001, Regression, Cox; The interim analysis only reported a p-value for testing whether the hazard ratio was not equal to 1.5

2. Primary Outcome: Complete Remission
Time Frame: After induction therapy was completed (1 or 2 months)
Population: Eligible patients who did not withdraw consent
Measure: Number; unit: participants
Groups:
- Ara-C+Daunomycin: A 21 day treatment cycle of Induction 7+3 with a 2nd 21 day cycle of the same for patients who did not achieve a complete remission during the first cycle of treatment
- Ara-C+Daunomycin+Mylotarg: A 21 day treatment cycle of Induction 7+3+G.O. with a 2nd 21 day cycle of the same for patients who did not achieve a complete remission (CR) during the first cycle of treatment
Arm/Group | Ara-C+Daunomycin | Ara-C+Daunomycin+Mylotarg
Number analyzed (Participants) | 296 | 300
participants | 203 | 207
Statistical Analysis 1: Comparison: Ara-C+Daunomycin vs Ara-C+Daunomycin+Mylotarg; Interim futility analysis alternative hypothesis based on the design specification that the 7+3+GO arm would have a 12% increase in CR rate; Test type: Superiority or Other; p < 0.0025, Test of difference of proportions

3. Secondary Outcome: Toxicity
Description: Number of patients with Grade 3-5 adverse events that are related to study drug by given type of adverse event
Time Frame: For induction, daily for the first 10 days, then twice weekly until consolidation treatment. Weekly during consolidation treatment. Weekly if randomized to post-consolidation G.O.
Population: Eligible patients who started therapy
Measure: Number; unit: Participants with a given type of AE
Groups:
- Ara-C Consolidation: For patients who achieved a CR during induction, patients may receive up to 3 28 day cycles of treatment with Ara-C consolidation. Patients who relapse from CR are taken off protocol consolidation treatment.
- Post-consolidation G.O.: For patients who remain in CR without relapse, patients may receive up to 3 doses of G.O. 28 days apart.
Arm/Group | Ara-C+Daunomycin+Mylotarg | Ara-C+Daunomycin | Ara-C Consolidation | Post-consolidation G.O.
Number analyzed (Participants) | 293 | 294 | 377 | 79
Participants with a given type of AE
  ALT, SGPT (serum glutamic pyruvic transaminase) | 29 | 11 | 22 | 2
  AST, SGOT (serum glut. oxaloacetic transaminase) | 32 | 11 | 17 | 2
  Acidosis (metabolic or respiratory) | 2 | 0 | 2 | 0
  Adult respiratory distress syndrome (ARDS) | 7 | 0 | 2 | 0
  Albumin, serum-low (hypoalbuminemia) | 15 | 10 | 3 | 0
  Alkaline phosphatase | 3 | 2 | 2 | 0
  Alkalosis (metabolic or respiratory) | 1 | 1 | 0 | 0
  Allergic reaction/hypersens. (inc drug fever) | 6 | 0 | 0 | 0
  Amylase | 0 | 0 | 1 | 0
  Anorexia | 14 | 13 | 2 | 0
  Apnea | 0 | 0 | 1 | 0
  Ataxia (incoordination) | 0 | 0 | 2 | 0
  Bicarbonate, serum-low | 1 | 0 | 0 | 0
  Bilirubin (hyperbilirubinemia) | 14 | 11 | 4 | 0
  Blood/Bone Marrow-Other (Specify) | 0 | 1 | 2 | 0
  Bronchospasm, wheezing | 1 | 0 | 0 | 0
  Calcium, serum-low (hypocalcemia) | 13 | 7 | 3 | 0
  Cardiac Arrhythmia-Other (Specify) | 0 | 0 | 1 | 0
  Cardiac General-Other (Specify) | 0 | 2 | 0 | 0
  Cardiac troponin I (cTnI) | 0 | 1 | 0 | 0
  Cardiac troponin T (cTnT) | 0 | 0 | 3 | 0
  Cardiac-ischemia/infarction | 2 | 1 | 4 | 0
  Colitis | 2 | 6 | 1 | 0
  Colitis, infectious (e.g., Clostridium difficile) | 8 | 10 | 4 | 0
  Confusion | 3 | 1 | 0 | 0
  Constipation | 1 | 0 | 0 | 0
  Cough | 0 | 0 | 1 | 0
  Creatinine | 3 | 2 | 0 | 0
  DIC (disseminated intravascular coagulation) | 2 | 0 | 0 | 0
  Death not assoc with CTCAE term-Multi-organ failu | 1 | 0 | 0 | 0
  Dehydration | 0 | 0 | 1 | 1
  Diarrhea | 5 | 19 | 4 | 0
  Distention/bloating, abdominal | 0 | 0 | 1 | 0
  Dizziness | 2 | 0 | 3 | 0
  Dysphagia (difficulty swallowing) | 1 | 1 | 0 | 0
  Dyspnea (shortness of breath) | 10 | 6 | 10 | 0
  Edema, larynx | 1 | 1 | 0 | 0
  Edema: limb | 0 | 0 | 1 | 0
  Edema: viscera | 1 | 0 | 0 | 0
  Enteritis (inflammation of the small bowel) | 1 | 0 | 0 | 0
  Esophagitis | 1 | 3 | 0 | 0
  Fatigue (asthenia, lethargy, malaise) | 24 | 25 | 22 | 4
  Febrile neutropenia | 178 | 196 | 183 | 22
  Fever (in the absence of neutropenia) | 6 | 8 | 16 | 1
  Fistula, GI - Rectum | 1 | 0 | 0 | 0
  Fistula, GU - Vagina | 1 | 0 | 0 | 0
  Flu-like syndrome | 0 | 0 | 1 | 0
  GGT (gamma-glutamyl transpeptidase) | 1 | 0 | 4 | 0
  Glucose, serum-high (hyperglycemia) | 22 | 12 | 15 | 2
  Glucose, serum-low (hypoglycemia) | 1 | 0 | 0 | 0
  Hematoma | 1 | 1 | 1 | 0
  Hemoglobin | 101 | 87 | 144 | 2
  Hemolysis | 0 | 0 | 1 | 0
  Hemorrhage, CNS | 5 | 1 | 0 | 0
  Hemorrhage, GI - Abdomen NOS | 0 | 1 | 0 | 0
  Hemorrhage, GI - Jejunum | 1 | 0 | 0 | 0
  Hemorrhage, GI - Lower GI NOS | 0 | 0 | 1 | 0
  Hemorrhage, GI - Oral cavity | 1 | 0 | 2 | 0
  Hemorrhage, GI - Rectum | 1 | 1 | 0 | 0
  Hemorrhage, GU - Bladder | 2 | 0 | 0 | 0
  Hemorrhage, GU - Kidney | 1 | 0 | 0 | 0
  Hemorrhage, GU - Urinary NOS | 1 | 0 | 0 | 0
  Hemorrhage, GU - Uterus | 0 | 2 | 0 | 0
  Hemorrhage, GU - Vagina | 1 | 1 | 1 | 0
  Hemorrhage, pulmonary/upper respiratory - Lung | 5 | 0 | 0 | 0
  Hemorrhage, pulmonary/upper respiratory - Nose | 3 | 1 | 4 | 0
  Hemorrhage/Bleeding-Other (Specify) | 8 | 5 | 12 | 0
  Hepatobiliary/Pancreas-Other (Specify) | 3 | 0 | 0 | 0
  Hiccoughs (hiccups, singultus) | 0 | 1 | 0 | 0
  Hypertension | 2 | 3 | 2 | 0
  Hypotension | 5 | 1 | 4 | 1
  Hypoxia | 8 | 2 | 6 | 0
  Infec with Grade 3 or 4 neut - Abdomen NOS | 1 | 0 | 0 | 0
  Infec with Grade 3 or 4 neut - Anal/perianal | 0 | 2 | 4 | 0
  Infec with Grade 3 or 4 neut - Appendix | 0 | 1 | 0 | 0
  Infec with Grade 3 or 4 neut - Bladder (urin | 2 | 1 | 4 | 0
  Infec with Grade 3 or 4 neut - Blood | 30 | 25 | 47 | 4
  Infec with Grade 3 or 4 neut - Bone (osteomy | 0 | 0 | 1 | 0
  Infec with Grade 3 or 4 neut - Brain + Spina | 0 | 1 | 0 | 0
  Infec with Grade 3 or 4 neut - Bronchus | 0 | 1 | 1 | 0
  Infec with Grade 3 or 4 neut - Catheter-rela | 5 | 6 | 13 | 2
  Infec with Grade 3 or 4 neut - Cecum | 0 | 0 | 1 | 0
  Infec with Grade 3 or 4 neut - Colon | 5 | 2 | 2 | 0
  Infec with Grade 3 or 4 neut - Dental-tooth | 1 | 2 | 3 | 0
  Infec with Grade 3 or 4 neut - Heart (endoca | 1 | 1 | 0 | 0
  Infec with Grade 3 or 4 neut - Lip/perioral | 1 | 0 | 0 | 0
  Infec with Grade 3 or 4 neut - Liver | 0 | 1 | 1 | 0
  Infec with Grade 3 or 4 neut - Lung (pneumon | 22 | 27 | 22 | 0
  Infec with Grade 3 or 4 neut - Meninges (men | 0 | 0 | 1 | 0
  Infect with Grade 3 or 4 neut - Mucosa | 1 | 2 | 1 | 0
  Infec with Grade 3 or 4 neut - Nerve-periphe | 1 | 0 | 0 | 0
  Infec with Grade 3 or 4 neut - Oral cavity-g | 2 | 3 | 2 | 0
  Infec with Grade 3 or 4 neut - Pelvis NOS | 1 | 0 | 0 | 0
  Infec with Grade 3 or 4 neut- Pharynx | 0 | 1 | 1 | 1
  Infec with Grade 3 or 4 neut - Rectum | 0 | 1 | 0 | 0
  Infec with Grade 3 or 4 neut - Sinus | 2 | 3 | 2 | 0
  Infec with Grade 3 or 4 neut - Skin (celluli | 4 | 3 | 9 | 1
  Infec with Grade 3 or 4 neut - Small bowel N | 0 | 1 | 1 | 0
  Infec with Grade 3 or 4 neut - Upper airway | 1 | 0 | 0 | 0
  Infection with Grade 3 or 4 neut - Urinary tract | 6 | 6 | 6 | 0
  Infec with Grade 3 or 4 neut - Vulva | 0 | 0 | 1 | 0
  Infec with Grade 3 or 4 neut - Wound | 1 | 0 | 0 | 0
  Infec with normal ANC or Grade 1/2 neut - Blood | 0 | 0 | 6 | 0
  Infec with norm ANC or Gr 1/2 neut, Catheter-rel | 0 | 1 | 4 | 0
  Infec with norm ANC or Grade 1/2 neut - Colon | 0 | 0 | 1 | 0
  Infec with norm ANC or Gr 1/2 neutr- Dental-tooth | 1 | 0 | 0 | 0
  Infec with norm ANC or Gr 1/2 neut - Heart | 0 | 0 | 1 | 0
  Infec with norm ANC or Gr 1/2 neutrophils - Liver | 1 | 0 | 0 | 0
  Infec with norm ANC or Gr 1/2 neut-Lung (pneumoni) | 6 | 0 | 9 | 0
  Infec with norm ANC or Gr 1/2 neut - Muscle | 1 | 0 | 0 | 0
  Inf with norm ANC or Gr 1/2 neut-Oral cavity-gums | 0 | 1 | 0 | 0
  Infec with norm ANC or Gr 1/2 neut - Scrotum | 0 | 0 | 1 | 0
  Infec with norm ANC or Gr 1/2 neut-Skin | 2 | 0 | 0 | 0
  Infec with norm ANC or Gr 1/2 neut-Urinary tract | 0 | 1 | 0 | 0
  Infection with unknown ANC - Blood | 0 | 3 | 7 | 0
  Infection with unknown ANC - Catheter-related | 3 | 1 | 1 | 0
  Infection with unknown ANC - Dental-tooth | 0 | 1 | 0 | 0
  Infection with unknown ANC - Joint | 0 | 0 | 2 | 0
  Infection with unknown ANC - Liver | 0 | 0 | 1 | 0
  Infection with unknown ANC - Lung (pneumonia) | 0 | 2 | 2 | 0
  Infection with unknown ANC - Mucosa | 0 | 0 | 1 | 0
  Infection with unknown ANC - Sinus | 1 | 1 | 0 | 0
  Infection with unknown ANC - Skin (cellulitis) | 4 | 3 | 3 | 0
  Infection with unknown ANC - Urinary tract NOS | 1 | 1 | 0 | 0
  Infection with unknown ANC - Wound | 0 | 1 | 0 | 0
  Infection-Other (Specify) | 4 | 4 | 4 | 0
  Left ventricular diastolic dysfunction | 0 | 0 | 1 | 0
  Left ventricular systolic dysfunction | 1 | 1 | 2 | 0
  Leukocytes (total WBC) | 106 | 96 | 151 | 41
  Leukoencephalopathy (radiolographic findings) | 0 | 0 | 1 | 0
  Liver dysfunction/failure (clinical) | 4 | 1 | 0 | 0
  Lymphopenia | 21 | 23 | 50 | 4
  Magnesium, serum-low (hypomagnesemia) | 1 | 1 | 1 | 0
  Metabolic/Laboratory-Other (Specify) | 3 | 5 | 4 | 0
  Mood alteration - anxiety | 1 | 0 | 1 | 0
  Mood alteration - depression | 0 | 1 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Esophagus | 0 | 1 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Large bowel | 0 | 1 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Larynx | 0 | 1 | 0 | 0
  Mucositis/stomatitis (clinical exam) - Oral cavity | 6 | 11 | 2 | 0
  Mucositis/stomatitis (clinical exam) - Pharynx | 2 | 2 | 0 | 0
  Mucositis/stomatitis (func/sympt) - Esophagus | 0 | 2 | 0 | 0
  Mucositis/stomatitis (func/sympt)- Oral cavity | 4 | 9 | 1 | 0
  Mucositis/stomatitis (func/sympt) - Pharynx | 1 | 2 | 1 | 0
  Muscle weakness (func/sym, Whole body/generalized | 0 | 1 | 2 | 0
  Nasal cavity/paranasal sinus reactions | 1 | 0 | 0 | 0
  Nausea | 7 | 13 | 7 | 1
  Necrosis, GI - Rectum | 0 | 0 | 1 | 0
  Neurology-Other (Specify) | 1 | 1 | 1 | 0
  Neuropathy: motor | 0 | 0 | 2 | 0
  Neuropathy: sensory | 1 | 0 | 1 | 0
  Neutrophils/granulocytes (ANC/AGC) | 111 | 110 | 193 | 43
  Nystagmus | 0 | 1 | 0 | 0
  Obstruction/stenosis of airway - Trachea | 0 | 0 | 1 | 0
  Ocular/Visual-Other (Specify) | 0 | 1 | 0 | 0
  Opportunistic infec assoc with Gr 2 lymphopenia | 0 | 2 | 0 | 1
  PTT (Partial thromboplastin time) | 0 | 0 | 1 | 0
  Pain - Abdomen NOS | 8 | 5 | 3 | 0
  Pain - Anus | 0 | 0 | 1 | 1
  Pain - Back | 1 | 0 | 1 | 1
  Pain - Bone | 0 | 0 | 4 | 0
  Pain - Chest/thorax NOS | 2 | 1 | 2 | 0
  Pain - Extremity-limb | 0 | 1 | 1 | 1
  Pain - Eye | 0 | 0 | 1 | 0
  Pain - Head/headache | 8 | 1 | 8 | 1
  Pain - Joint | 1 | 0 | 0 | 0
  Pain - Muscle | 0 | 0 | 1 | 0
  Pain - Oral-gums | 0 | 1 | 0 | 0
  Pain - Rectum | 0 | 0 | 0 | 1
  Pain - Throat/pharynx/larynx | 0 | 1 | 0 | 0
  Pain-Other (Specify) | 1 | 0 | 0 | 0
  Pancreatic endocrine: glucose intolerance | 1 | 0 | 0 | 0
  Perforation, GI - Colon | 0 | 1 | 0 | 0
  Pericardial effusion (non-malignant) | 1 | 0 | 0 | 0
  Pericarditis | 1 | 0 | 0 | 0
  Petechiae/purpura | 6 | 2 | 3 | 1
  Phosphate, serum-low (hypophosphatemia) | 10 | 9 | 6 | 1
  Platelets | 145 | 130 | 226 | 40
  Pleural effusion (non-malignant) | 1 | 1 | 3 | 0
  Pneumonitis/pulmonary infiltrates | 3 | 1 | 5 | 0
  Portal vein flow | 2 | 0 | 0 | 0
  Potassium, serum-high (hyperkalemia) | 4 | 2 | 0 | 0
  Potassium, serum-low (hypokalemia) | 21 | 15 | 19 | 3
  Proctitis | 0 | 1 | 0 | 0
  Pulmonary/Upper Respiratory-Other (Specify) | 1 | 0 | 1 | 0
  Rash/desquamation | 6 | 9 | 1 | 0
  Renal failure | 8 | 6 | 0 | 0
  Rigors/chills | 0 | 0 | 1 | 0
  Seroma | 1 | 0 | 0 | 0
  Serum sickness | 0 | 0 | 0 | 1
  Sodium, serum-high (hypernatremia) | 2 | 0 | 0 | 0
  Sodium, serum-low (hyponatremia) | 8 | 15 | 4 | 0
  Somnolence/depressed level of consciousness | 1 | 0 | 0 | 0
  Atrial fibrillation | 0 | 1 | 0 | 0
  Sinus tachycardia | 1 | 0 | 0 | 0
  Supraventricular arrhythmia NOS | 1 | 0 | 0 | 0
  Syncope (fainting) | 1 | 3 | 4 | 0
  Syndromes-Other (Specify) | 0 | 0 | 2 | 0
  Thrombosis/embolism (vascular access-related) | 0 | 1 | 1 | 0
  Thrombosis/thrombus/embolism | 4 | 4 | 4 | 0
  Thrombotic microangiopathy | 0 | 1 | 0 | 0
  Tumor lysis syndrome | 2 | 2 | 0 | 0
  Typhlitis (cecal inflammation) | 3 | 4 | 1 | 0
  Uric acid, serum-high (hyperuricemia) | 1 | 0 | 1 | 0
  Vasovagal episode | 0 | 0 | 1 | 0
  Ventricular arrhythmia - Ventricular fibrillation | 1 | 0 | 0 | 0
  Vision-blurred vision | 0 | 1 | 0 | 0
  Vomiting | 2 | 5 | 5 | 1

ADVERSE EVENTS:
Time Frame: While the patient is on treatment until resolution of acute toxicities with maximum grade reported.
Description: Regular investigator assessments are reported after each cycle of protocol treatment.
Groups:
- Induction 7 + 3 + G.O.: A 21 day treatment cycle of Induction 7+3+G.O. with a 2nd 21 day cycle of the same for patients who did not achieve a complete remission (CR) during the first cycle of treatment
- Induction 7 + 3: A 21 day treatment cycle of Induction 7+3 with a 2nd 21 day cycle of the same for patients who did not achieve a complete remission during the first cycle of treatment
Arm/Group | Induction 7 + 3 + G.O. | Induction 7 + 3 | Ara-C Consolidation | Post-consolidation G.O.
Serious Adverse Events (participants affected / at risk) | 47/293 | 9/293 | 13/375 | 19/78
Other Adverse Events (participants affected / at risk) | 277/293 | 279/293 | 356/375 | 77/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction 7 + 3 + G.O. (N=293) | Induction 7 + 3 (N=293) | Ara-C Consolidation (N=375) | Post-consolidation G.O. (N=78)
DIC (disseminated intravascular coagulation) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 1 (1) | 4 (4) | 9 (9)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac-ischemia/infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain - Rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perforation, GI - Colon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death not associated with CTCAE term - Multi-organ failure (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syndromes-Other (Specify) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary/Pancreas-Other (Specify) (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Portal vein flow (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 8 (8) | 2 (2) | 1 (1) | 3 (3)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Colon (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Heart (endoca (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (pneumon (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Pelvis NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Skin (celluli (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infection-Other (Specify) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 5 (5) | 0 (0) | 1 (1) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Alkaline phosphatase (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Creatinine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytes (total WBC) (Investigations) | 5 (5) | 0 (0) | 1 (1) | 2 (2)
Metabolic/Laboratory-Other (Specify) (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3 (3) | 0 (0) | 1 (1) | 5 (5)
Platelets (Investigations) | 9 (9) | 1 (1) | 1 (1) | 2 (2)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic endocrine: glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, CNS (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (radiolographic findings) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurology-Other (Specify) (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GU - Bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, GU - Kidney (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemorrhage/Bleeding-Other (Specify) (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction 7 + 3 + G.O. (N=293) | Induction 7 + 3 (N=293) | Ara-C Consolidation (N=375) | Post-consolidation G.O. (N=78)
Febrile neutropenia (Blood and lymphatic system disorders) | 172 (172) | 194 (194) | 178 (178) | 14 (14)
Hemoglobin (Blood and lymphatic system disorders) | 116 (116) | 109 (109) | 201 (201) | 27 (27)
Vision-blurred vision (Eye disorders) | 0 (0) | 0 (0) | 19 (19) | 0 (0)
Constipation (Gastrointestinal disorders) | 36 (36) | 32 (32) | 46 (46) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 115 (115) | 130 (130) | 76 (76) | 9 (9)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 25 (25) | 20 (20) | 0 (0)
Hemorrhage, GI - Oral cavity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 19 (19) | 0 (0)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 76 (76) | 64 (64) | 63 (63) | 8 (8)
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 33 (33) | 37 (37) | 35 (35) | 0 (0)
Nausea (Gastrointestinal disorders) | 165 (165) | 159 (159) | 182 (182) | 40 (40)
Pain - Abdomen NOS (Gastrointestinal disorders) | 51 (51) | 35 (35) | 31 (31) | 8 (8)
Vomiting (Gastrointestinal disorders) | 93 (93) | 75 (75) | 97 (97) | 22 (22)
Edema: limb (General disorders) | 38 (38) | 24 (24) | 27 (27) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 140 (140) | 142 (142) | 210 (210) | 41 (41)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC lt1.0 x 10e9/L) (General disorders) | 56 (56) | 55 (55) | 97 (97) | 14 (14)
Rigors/chills (General disorders) | 71 (71) | 55 (55) | 56 (56) | 8 (8)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 15 (15) | 0 (0) | 0 (0) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Blood (Infections and infestations) | 23 (23) | 24 (24) | 47 (47) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Lung (pneumon (Infections and infestations) | 22 (22) | 26 (26) | 23 (23) | 0 (0)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 124 (124) | 90 (90) | 137 (137) | 34 (34)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 126 (126) | 92 (92) | 121 (121) | 33 (33)
Alkaline phosphatase (Investigations) | 79 (79) | 60 (60) | 84 (84) | 22 (22)
Bilirubin (hyperbilirubinemia) (Investigations) | 51 (51) | 63 (63) | 75 (75) | 0 (0)
Creatinine (Investigations) | 34 (34) | 19 (19) | 23 (23) | 0 (0)
Leukocytes (total WBC) (Investigations) | 101 (101) | 97 (97) | 152 (152) | 40 (40)
Lymphopenia (Investigations) | 32 (32) | 27 (27) | 50 (50) | 10 (10)
Metabolic/Laboratory-Other (Specify) (Investigations) | 16 (16) | 0 (0) | 21 (21) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 109 (109) | 111 (111) | 195 (195) | 40 (40)
Platelets (Investigations) | 136 (136) | 130 (130) | 227 (227) | 49 (49)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 69 (69) | 53 (53) | 81 (81) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 85 (85) | 75 (75) | 76 (76) | 9 (9)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 44 (44) | 53 (53) | 44 (44) | 5 (5)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 79 (79) | 71 (71) | 97 (97) | 21 (21)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 17 (17) | 0 (0) | 25 (25) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 17 (17) | 18 (18) | 0 (0) | 0 (0)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 20 (20) | 0 (0) | 0 (0) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 55 (55) | 44 (44) | 61 (61) | 12 (12)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 42 (42) | 41 (41) | 39 (39) | 8 (8)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 20 (20) | 0 (0)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 15 (15) | 40 (40) | 8 (8)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 21 (21) | 4 (4)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 19 (19) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 42 (42) | 0 (0)
Pain - Head/headache (Nervous system disorders) | 72 (72) | 48 (48) | 94 (94) | 9 (9)
Taste alteration (dysgeusia) (Nervous system disorders) | 18 (18) | 16 (16) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 25 (25) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 0 (0) | 20 (20) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 33 (33) | 20 (20) | 59 (59) | 0 (0)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 37 (37) | 24 (24) | 26 (26) | 6 (6)
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 76 (76) | 98 (98) | 118 (118) | 8 (8)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 53 (53) | 45 (45) | 85 (85) | 0 (0)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 15 (15) | 20 (20) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 51 (51) | 64 (64) | 62 (62) | 6 (6)
Hemorrhage/Bleeding-Other (Specify) (Vascular disorders) | 27 (27) | 15 (15) | 29 (29) | 0 (0)
Hypertension (Vascular disorders) | 21 (21) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 17 (17) | 15 (15) | 28 (28) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No